CLINICAL TRIAL: NCT00300079
Title: A Multiple-Dose Study of the IOP-Lowering Efficacy of Azopt 1.0% Compared to Timolol 0.5% When Added to a PGA as Adjunctive Therapy Over a 24 Hour Period in Patients With Glaucoma or Ocular Hypertension
Brief Title: Study of the Intraocular Pressure (IOP)-Lowering Efficacy of Azopt 1.0% Compared to Timolol 0.5% in Patients With Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Collaborators: University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CM-05-13; CM-05-13
Record Dates: First submitted 2006-03-06; First posted 2006-03-08 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2008-06

CONDITIONS: Primary Open Angle Glaucoma; Ocular Hypertension
Keywords: Ocular Hypertension Patients
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

INTERVENTIONS:
Drug: brinzolamide 1.0%

SUMMARY:
This is a multiple-dose study of the IOP-lowering efficacy of Azopt (brinzolamide) 1.0% compared to timolol 0.5% when added to a prostaglandin analogue (PGA) as adjunctive therapy over a 24 hour period in patients with glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Primary open angle glaucoma or ocular hypertension patients

Exclusion Criteria:

* Women of childbearing potential
* History of bronchial asthma, or severe chronic obstructive pulmonary disease
* Presence of acute glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-09; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
IOP-lowering at 8 and 16 weeks

SECONDARY OUTCOMES:
Safety throughout the 16 weeks of the study

CONTACTS AND LOCATIONS:
Overall Officials: John Liu, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- San Diego, California, United States

REFERENCES:
- [Result] Liu JH, Medeiros FA, Slight JR, Weinreb RN. Comparing diurnal and nocturnal effects of brinzolamide and timolol on intraocular pressure in patients receiving latanoprost monotherapy. Ophthalmology. 2009 Mar;116(3):449-54. doi: 10.1016/j.ophtha.2008.09.054. Epub 2009 Jan 20. PMID 19157559